CLINICAL TRIAL: NCT01221350
Title: Exploratory Study of Lipoic Acid Supplementation on Oxidative Stress, Inflammatory and Functional Markers in Asthmatic Patients: Randomized, Double-Blind, Placebo-Controlled, Parallel-Group Clinical Trial.
Brief Title: Effects of Lipoic Acid on Oxidative, Inflammatory and Functional Markers in Asthmatic Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centro Universitario de Ciencias de la Salud, Mexico (Other)
Collaborators: National Council of Science and Technology, Mexico (Other); University of Guadalajara (Other); Hospital Civil Juan I. Menchaca (Other)
Responsible Party: Principal Investigator, Fernando Siller-Lopez, Research professor, Centro Universitario de Ciencias de la Salud, Mexico
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: UdeG-FSL-2010; Salud-2010-C01-140590 (Other Grant/Funding Number: Fondo Sectorial de Investigación en Salud, Conacyt)
Record Dates: First submitted 2010-10-14; First posted 2010-10-15 (Estimated); Results first posted 2013-07-30 (Estimated); Last update posted 2013-11-08 (Estimated); Status verified 2013-10

CONDITIONS: Asthma; Allergic Rhinitis
Keywords: Asthma; Allergic rhinitis; Respiratory disease; Allergy; Lipoic acid; Thioctic acid; Antioxidant; Oxidative stress
MeSH Terms: conditions — Asthma; Rhinitis, Allergic; Respiration Disorders; Hypersensitivity | interventions — Thioctic Acid; Placebo Effect

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lipoic acid (Experimental): Lipoic acid 600 mg oral dose (two 300 mg capsules) once daily in the morning during 60 days
  Interventions: Dietary Supplement: Lipoic acid
- Placebo (Placebo Comparator): Placebo (two placebo capsules) orally once daily in the morning during 60 days
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Lipoic acid — Lipoic acid 600 mg dose (two 300 mg capsules) once daily in the morning. All patients continued their asthma treatments given by their primary care physician also they were allowed to use rescue medication on demand consisting in inhaled salbutamol. During basal and 8 weeks visits spirometry with bronchodilator challenge, sputum induction and quality of life questionnaires and asthma control test were performed.
  Other Names: Thioctic Acid; Alpha-Lipoic Acid
  Arms: Lipoic acid
Dietary Supplement: Placebo — Placebo (two capsules filled with 300 mg vehicle) once daily in the morning during 60 days. All patients continued their asthma treatments given by their primary care physician also they were allowed to use rescue medication on demand consisting in inhaled salbutamol. During basal and 8 weeks visits spirometry with bronchodilator challenge, sputum induction and quality of life questionnaires and asthma control test were performed
  Other Names: Placebos; Placebo effect
  Arms: Placebo

SUMMARY:
The aim of the study is to use the antioxidant and antiinflammatory effects of lipoic acid to improve the quality of life of patients with asthma.

The investigators will administrate 600 mg lipoic acid orally on a daily basis during two months concurrent with the patient anti-asthmatic therapy and evaluate the effects on resulting pulmonary function, inflammatory and oxidative stress biomarkers and health-related quality of life previous to the initial of the treatment and at 60 days of the supplementary therapy.

DETAILED DESCRIPTION:
Asthma is an inflammatory disease of high prevalence around the world. During development of asthma the presence of oxidative stress has been related to susceptibility and severity of the disease, thus making the use of antioxidant adjuvant therapy with lipoic acid (LA) an interesting treatment option. The objective of the study is to evaluate the efficacy of LA as an adjuvant treatment on functional, antioxidant, inflammatory, quality and control parameters of asthma in human subjects. The trial design is a randomized, double blind, placebo controlled parallel study.

Adult patients (>18 years) with history of mild intermittent to moderate asthma according to the Global Initiative for Asthma (GINA) guidelines were enrolled. It was required a positive skin prick test (>3 mm) for at least two regional allergens. Patients were randomly assigned to receive lipoic acid or placebo for 60 days. Participants had an intermediate visit to the attending physician one month after initial of treatment to monitor adverse events and to undergo laboratory tests.

1. Introduction. Asthma is an inflammatory disease of high prevalence around the world. During development of asthma the presence of oxidative stress has been related to susceptibility and severity of the disease, thus making the use of antioxidant adjuvant therapy with lipoic acid (LA) an interesting treatment option.
2. Study design. A randomized, double blind, placebo controlled parallel study
3. Methods. Participants and interventions: 55 patients with mild to moderate asthma from Hospital Civil "Juan I. Menchaca" in Guadalajara, Jalisco, México were included and randomized in block of 10 to receive; LA (600 mg/day) or placebo for eight weeks from January to October of 2011.
4. Objective. To evaluate the efficacy of LA as an adjuvant treatment on functional, antioxidant, inflammatory, quality and control parameters of asthma in human subjects. Primary outcome: change on Forced expiratory volume in 1 second (FEV1), secondary outcomes were levels of Oxygen radical absorbance capacity (ORAC), glutathione (GSH), glutathione disulfide (GSSG), protein carbonyls, differential count of sputum cells, interleukin-4 (IL-4) and scores of quality of life and control of asthma questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Outpatients (≥18 and ≤ 75 years of age) female or male
* Willingness to participate and comply with procedures by signing a written informed consent
* Moderate/severe persistent allergic rhinitis according to Allergic Rhinitis and its Impact on Asthma (ARIA) guidelines with a history of intermittent, mild persistent or moderate persistent asthma according to GINA guidelines
* Confirmed allergy to at least one of the following allergen preparations: house dust mite f; house dust mite p; cockroach; bush mix; tree mix; grass mix; weed mix, cat; or dog.
* All prior medication washout times had been observed
* Female volunteers of childbearing potential had to agree to use a medically accepted method of contraception
* Negative urine pregnancy test
* Without a concomitant chronic medical condition (e.g., significant cardiovascular disease, diabetes requiring medication, chronic kidney disease, chronic thyroid disease, or coagulation defects)
* Willingness to adhere to the dosing and visit schedules

Exclusion Criteria:

* Pregnant or breastfeeding
* Female who was or intended to become pregnant during the study or within 12 weeks after study completion
* Taking medications prohibited during the study or had not complied with the requirements for the designated washout periods for any of the prohibited medications
* Anatomical abnormalities of the nose (turbinate hypertrophy, septal deviation, polyps)
* Acute or chronic sinusitis currently being treated with antibiotics and/or topical or oral decongestants
* Upper respiratory tract or sinus infection that required antibiotic therapy and had not had at least a 14-day wash-out period prior to the run-in period
* Patients undergoing a progressive course of immunotherapy. Subjects on a regular maintenance schedule prior to the screening visit are eligible for study inclusion; however, subject could not receive hyposensitization treatment within 24 hours prior to any study visit
* Concomitant medical problem
* In a situation or condition that could interfere with participation in the study
* Allergic or sensitivity to the study drug or its excipients
* History of inadequate adherence to treatment

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2010-11; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Fernando R. Siller Lopez, PhD, Principal Investigator — Centro Universitario de Ciencias de la Salud, Mexico
Locations (2):
- Mexico (2):
  - Hospital Civil de Guadalajara "Juan I. Menchaca", Guadalajara, Jalisco
  - Departamento de Fisiología, CUCS, UdeG, Guadalajara, Jalisco

REFERENCES:
- [Background] Kroegel C. [Global Initiative for Asthma Management and Prevention--GINA 2006]. Pneumologie. 2007 May;61(5):295-304. doi: 10.1055/s-2007-959180. German. PMID 17523070
- [Background] Brozek JL, Bousquet J, Baena-Cagnani CE, Bonini S, Canonica GW, Casale TB, van Wijk RG, Ohta K, Zuberbier T, Schunemann HJ; Global Allergy and Asthma European Network; Grading of Recommendations Assessment, Development and Evaluation Working Group. Allergic Rhinitis and its Impact on Asthma (ARIA) guidelines: 2010 revision. J Allergy Clin Immunol. 2010 Sep;126(3):466-76. doi: 10.1016/j.jaci.2010.06.047. PMID 20816182
- [Background] Cho YS, Lee J, Lee TH, Lee EY, Lee KU, Park JY, Moon HB. alpha-Lipoic acid inhibits airway inflammation and hyperresponsiveness in a mouse model of asthma. J Allergy Clin Immunol. 2004 Aug;114(2):429-35. doi: 10.1016/j.jaci.2004.04.004. PMID 15316528
- [Background] Lee KS, Kim SR, Park SJ, Min KH, Lee KY, Jin SM, Yoo WH, Lee YC. Antioxidant down-regulates interleukin-18 expression in asthma. Mol Pharmacol. 2006 Oct;70(4):1184-93. doi: 10.1124/mol.106.024737. Epub 2006 Jul 5. PMID 16822930
- [Background] Patel BD, Welch AA, Bingham SA, Luben RN, Day NE, Khaw KT, Lomas DA, Wareham NJ. Dietary antioxidants and asthma in adults. Thorax. 2006 May;61(5):388-93. doi: 10.1136/thx.2004.024935. Epub 2006 Feb 7. PMID 16467075
- [Background] Miller AL. The etiologies, pathophysiology, and alternative/complementary treatment of asthma. Altern Med Rev. 2001 Feb;6(1):20-47. PMID 11207455
- [Background] Rahman I. Oxidative stress, chromatin remodeling and gene transcription in inflammation and chronic lung diseases. J Biochem Mol Biol. 2003 Jan 31;36(1):95-109. doi: 10.5483/bmbrep.2003.36.1.095. PMID 12542980
- [Background] Biewenga GP, Haenen GR, Bast A. The pharmacology of the antioxidant lipoic acid. Gen Pharmacol. 1997 Sep;29(3):315-31. doi: 10.1016/s0306-3623(96)00474-0. PMID 9378235
- [Background] Singh U, Jialal I. Alpha-lipoic acid supplementation and diabetes. Nutr Rev. 2008 Nov;66(11):646-57. doi: 10.1111/j.1753-4887.2008.00118.x. PMID 19019027 (Retraction: PMID 22835141 Nutr Rev. 2012 Aug;70(8):482)
- [Background] Juniper EF, Guyatt GH, Epstein RS, Ferrie PJ, Jaeschke R, Hiller TK. Evaluation of impairment of health related quality of life in asthma: development of a questionnaire for use in clinical trials. Thorax. 1992 Feb;47(2):76-83. doi: 10.1136/thx.47.2.76. PMID 1549827
- [Background] Schatz M, Sorkness CA, Li JT, Marcus P, Murray JJ, Nathan RA, Kosinski M, Pendergraft TB, Jhingran P. Asthma Control Test: reliability, validity, and responsiveness in patients not previously followed by asthma specialists. J Allergy Clin Immunol. 2006 Mar;117(3):549-56. doi: 10.1016/j.jaci.2006.01.011. PMID 16522452
- [Background] Riedl MA, Saxon A, Diaz-Sanchez D. Oral sulforaphane increases Phase II antioxidant enzymes in the human upper airway. Clin Immunol. 2009 Mar;130(3):244-51. doi: 10.1016/j.clim.2008.10.007. Epub 2008 Nov 22. PMID 19028145
- [Background] Comhair SA, Erzurum SC. Redox control of asthma: molecular mechanisms and therapeutic opportunities. Antioxid Redox Signal. 2010 Jan;12(1):93-124. doi: 10.1089/ars.2008.2425. PMID 19634987
- [Background] Shay KP, Moreau RF, Smith EJ, Smith AR, Hagen TM. Alpha-lipoic acid as a dietary supplement: molecular mechanisms and therapeutic potential. Biochim Biophys Acta. 2009 Oct;1790(10):1149-60. doi: 10.1016/j.bbagen.2009.07.026. Epub 2009 Aug 4. PMID 19664690
- See also: Health Sciences Center, University of Guadalajara — http://www.cucs.udg.mx
- See also: Hospital Civil de Guadalajara — http://www.hcg.udg.mx/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 82 adult patients (>18 years) with history of mild intermittent to moderate asthma according to the Global Initiative for Asthma (GINA) guidelines were screened to participate in the study. Recruitment period: January-September 2011.
Pre-assignment Details: 55 patients were enrolled in the study prior to randomization and group assignment. From the 82 patients initially screened, 12 patients declined to participate and 15 patients did not meet the inclusion criteria.
Groups:
- Lipoic Acid: Lipoic acid 600 mg dose (two 300 mg capsules, p.o) once daily in the morning
- Placebo: Placebo 600 mg vehicle (two 300 mg capsules, p.o) once daily in the morning
Period: Overall Study
Arm/Group | Lipoic Acid | Placebo
Started | 28 | 27
Received Intervention | 28 | 27
Analysis Population | 23 | 24
Completed | 23 | 24
Not Completed | 5 | 3
Not completed — Discontinued intervention (GERD) | 1 | 0
Not completed — Exclusion criteria, asthma exacerbation | 0 | 1
Not completed — Withdrawal by Subject | 4 | 2

BASELINE CHARACTERISTICS:
Population: Patients with asthma from the occidental region of Mexico
Groups:
- Lipoic Acid: Lipoic acid (ALA) 600 mg oral dose (two 300 mg capsules) once daily in the morning during 60 days
- Placebo: Placebo (two 300 mg capsules filled with vehicle) orally once daily in the morning during 60 days
- Total: Total of all reporting groups
Arm/Group | Lipoic Acid | Placebo | Total
Number analyzed (Participants) | 28 | 27 | 55
Age Continuous [Mean (Standard Deviation); unit: years] | 40.9 (10.5) | 43.8 (16.6) | 42.3 (13.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 15 | 31
  Male | 12 | 12 | 24
Region of Enrollment [Number; unit: participants]
  Mexico | 28 | 27 | 55
Weight [Mean (Standard Deviation); unit: Kg] | 73.6 (16.1) | 74.1 (15.9) | 73.8 (16.0)
Body mass index (BMI) [Mean (Standard Deviation); unit: Kg/m^2] | 29.9 (5.4) | 28.0 (5.0) | 29.0 (5.2)

OUTCOME MEASURES:

1. Primary Outcome: Spirometric FVC Values at Baseline
Description: Measurement of spirometric predicted parameters at baseline. Forced vital capacity (FVC) is the volume of air that can forcibly be blown out after full inspiration, measured in liters.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | Lipoic Acid | Placebo
Number analyzed (Participants) | 23 | 24
Liters | 2.74 (0.68) | 3.07 (0.76)

2. Secondary Outcome: Induced Sputum of Glutathione (GSH)/Glutathione Disulfide (GSSG) Ratio at Baseline
Description: Induced sputum of GSH and GSSG levels at baseline. The ratio GSH/GSSG is considered an index of antioxidant status and reductive -SH groups. GSH and GSSG were measured by a microplate fluorescent assay.
Time Frame: Baseline
Measure: Mean (95% Confidence Interval); unit: ratio
Arm/Group | Lipoic Acid | Placebo
Number analyzed (Participants) | 23 | 24
ratio | 81.42 [65.31 to 97.52] | 35.77 [11.57 to 39.9]

3. Secondary Outcome: Induced Sputum of Glutathione (GSH)/Glutathione Disulfide (GSSG) Ratio at Endpoint
Description: Change in the induced sputum of antioxidant parameters GSH and GSSG levels after 60 days of treatment. The ratio GSH/GSSG is considered an index of antioxidant status and reductive -SH groups. GSH and GSSG were measured by a microplate fluorescent assay.
Time Frame: 60 days
Measure: Mean (95% Confidence Interval); unit: ratio
Arm/Group | Lipoic Acid | Placebo
Number analyzed (Participants) | 23 | 24
ratio | 58.6 [29.9 to 77.2] | 37.5 [13.4 to 55.9]

4. Secondary Outcome: Induced Sputum Carbonylated Proteins at Baseline
Description: Proteins can become modified by a large number of reactions involving reactive oxygen species. Among these, carbonylation is an irreversible and unrepairable oxidative reaction. The main protein modifications originated from oxidative stress comprise direct oxidation of aminoacids with a thiol group, such as cysteine, oxidative glycation, and carbonylation. Oxidative protein carbonylation induce protein degradation in a nonspecific manner. Chemically, oxidative carbonylation preferentially occurs at proline, threonine, lysine, and arginine, presumably through a metal-catalyzed activation of hydrogen peroxide to a reactive intermediate. Carbonylation usually refers to a process that forms reactive ketones or aldehydes that can be reacted by 2,4-dinitrophenylhydrazine (DNPH) to form hydrazones. Direct oxidation of side chains of lysine, arginine, proline, and threonine residues, among other aminoacids, produces DNPH detectable protein products
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: nmol/mg
Arm/Group | Lipoic Acid | Placebo
Number analyzed (Participants) | 23 | 24
nmol/mg | 7.5 (4.37) | 10.12 (10.81)

5. Primary Outcome: Spirometric FVC Values at Endpoint
Description: Measurement of spirometric predicted parameters at the baseline and after 60 days of treatment: Forced vital capacity (FVC) is the volume of air that can forcibly be blown out after full inspiration, measured in liters.
Time Frame: 60 days
Population: Per protocol
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | Lipoic Acid | Placebo
Number analyzed (Participants) | 23 | 24
Liters | 2.82 (0.77) | 3.06 (0.71)

6. Secondary Outcome: Induced Sputum Carbonylated Proteins at Endpoint
Description: as for outcome 4
Time Frame: 60 days
Measure: Mean (Standard Deviation); unit: nmol/mg
Arm/Group | Lipoic Acid | Placebo
Number analyzed (Participants) | 23 | 24
nmol/mg | 3.24 (2.2) | 4.21 (2.47)

7. Primary Outcome: Spirometric FEV1 Values at Baseline
Description: Measurement of spirometric predicted parameters at baseline: Forced expiratory volume in 1 second (FEV1), volume that has been exhaled at the end of the first second of forced expiration.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | Lipoic Acid | Placebo
Number analyzed (Participants) | 23 | 24
Liters | 2.01 (0.63) | 2.37 (0.65)

8. Primary Outcome: Spirometric FEV1 Values at Endpoint
Description: Measurement of spirometric predicted parameters after 60 days of treatment. Forced expiratory volume in 1 second (FEV1), volume that has been exhaled at the end of the first second of forced expiration.
Time Frame: 60 days
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | Lipoic Acid | Placebo
Number analyzed (Participants) | 23 | 24
Liters | 2.26 (0.69) | 2.35 (0.66)

9. Primary Outcome: Spirometric FEF Values at Baseline
Description: Measurement of spirometric parameters at baseline: Forced expiratory flow (FEF) is the flow (or speed) of air coming out of the lung during the middle portion of a forced expiration.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: Liters/sec
Arm/Group | Lipoic Acid | Placebo
Number analyzed (Participants) | 23 | 24
Liters/sec | 4.89 (1.72) | 6.09 (1.96)

10. Primary Outcome: Spirometric FEF Values at Endpoint
Description: Measurement of spirometric FEF after 60 days of treatment: Forced expiratory flow (FEF) is the flow (or speed) of air coming out of the lung during the middle portion of a forced expiration.
Time Frame: 60 days
Measure: Mean (Standard Deviation); unit: Liters/sec
Arm/Group | Lipoic Acid | Placebo
Number analyzed (Participants) | 23 | 24
Liters/sec | 5.47 (1.53) | 6.10 (1.68)

11. Secondary Outcome: Induced Sputum Eosinophils at Baseline
Description: Eosinophils, a prominent feature of asthma, are found in increased numbers in the circulation and sputum, usually in relation to the severity of asthma.
Time Frame: Baseline
Measure: Mean (95% Confidence Interval); unit: Eosinophil percentage in sputum cells
Units Other Than Participants: Eosinophils content
Arm/Group | Lipoic Acid | Placebo
Number analyzed (Participants) | 23 | 24
Number analyzed (Eosinophils content) | 100 | 300
Eosinophil percentage in sputum cells | 12.88 [2.5 to 13.3] | 6.10 [1.85 to 8.25]

12. Secondary Outcome: Induced Sputum Eosinophils at Endpoint
Description: as for outcome 11
Time Frame: 60 days
Measure: Mean (95% Confidence Interval); unit: Eosinophil percentage in sputum cells
Units Other Than Participants: Eosinophils content
Arm/Group | Lipoic Acid | Placebo
Number analyzed (Participants) | 23 | 24
Number analyzed (Eosinophils content) | 100 | 300
Eosinophil percentage in sputum cells | 6.39 [0.8 to 7] | 5.68 [0.8 to 7.9]

13. Secondary Outcome: Inflammatory Interleukin-4 (IL-4) Sputum Levels at Baseline
Description: Inflammatory IL-4 sputum levels after 60 days of treatment. Sputum induction is a semi-invasive technique used to detect and monitor airway inflammation. IL-4 is a Th2 cytokine that promote airway inflammation in asthma. IL-4 drives the production of immunoglobulin E (IgE) in B cells. IL-4 was measured by ELISA.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Lipoic Acid | Placebo
Number analyzed (Participants) | 23 | 24
pg/mL | 37.77 (38.04) | 39.90 (50.03)

14. Secondary Outcome: Inflammatory IL-4 Sputum Levels at Endpoint
Description: Inflammatory IL-4 sputum levels after 60 days of treatment. Sputum induction is a semi-invasive technique used to detect and monitor airway inflammation. IL-4 is a Th2 cytokine that promote airway inflammation in asthma. IL-4 drives the production of IgE in B cells. IL-4 was measured by ELISA.
Time Frame: 60 days
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Lipoic Acid | Placebo
Number analyzed (Participants) | 23 | 24
pg/mL | 14.53 (12.96) | 23.19 (34.39)

15. Secondary Outcome: Measurement of Quality of Life With the ACT (Asthma Control Test) at Baseline
Description: Assessment of Quality of life scores with the ACT (Asthma Control Test). The ACT is a way to determine if the asthma symptoms are well controlled. The Asthma Control Test™ (ACT™) is a five question health survey used to measure asthma control in individuals 12 years of age and older. The survey measures the elements of asthma control as defined by the National Heart, Lung, and Blood Institute (NHLBI). ACT is an efficient, reliable, and valid method of measuring asthma control, with or without, lung functioning measures such as spirometry. Each item includes 5 response options corresponding to a 5-point Likert-type rating scale. In scoring the ACT survey, responses for each of the 5 items are summed to yield a score ranging from 5 (poor control of asthma) to 25 (complete control of asthma).
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lipoic Acid | Placebo
Number analyzed (Participants) | 23 | 24
units on a scale | 13.65 (4.35) | 14.46 (4.85)

16. Secondary Outcome: Measurement of Quality of Life With the ACT (Asthma Control Test) at Endpoint
Description: as for outcome 15
Time Frame: 60 days
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lipoic Acid | Placebo
Number analyzed (Participants) | 23 | 24
units on a scale | 19.13 (3.62) | 17.71 (4.03)

17. Secondary Outcome: Measurement of Quality of Life With the AQLQ (Asthma Quality of Life Questionnaire) at Baseline
Description: The Asthma Quality of Life Questionnaire (AQLQ) was developed to measure the functional problems (physical, emotional, social and occupational) that are most troublesome to adults (17-70 years) with asthma.
  There are 32 questions in the AQLQ and they are in 4 domains (symptoms, activity limitation, emotional function and environmental stimuli). The activity domain contains 5 'patient-specific' questions. This allows patients to select 5 activities in which they are most limited and these activities will be assessed at each follow-up. Patients are asked to think about how they have been during the previous two weeks and to respond to each of the 32 questions on a 7-point scale (7 = not impaired at all - 1 = severely impaired). The overall AQLQ score is the mean of all 32 responses and the individual domain scores are the means of the items in those domains (http://www.qoltech.co.uk/aqlq.html).
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lipoic Acid | Placebo
Number analyzed (Participants) | 23 | 24
units on a scale | 3.86 (1.32) | 3.72 (1.61)

18. Secondary Outcome: Measurement of Quality of Life With the AQLQ (Asthma Quality of Life Questionnaire) at Endpoint
Description: as for outcome 17
Time Frame: 60 days
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lipoic Acid | Placebo
Number analyzed (Participants) | 23 | 24
units on a scale | 5.57 (1.17) | 5.10 (1.24)

ADVERSE EVENTS:
Time Frame: 60 days
Description: Serious or Other (non-serious) Adverse Events were collected/assessed, but none were observed during the 60 days period of intervention.
Arm/Group | Lipoic Acid | Placebo
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/24
Other Adverse Events (participants affected / at risk) | 0/23 | 0/24

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No